CLINICAL TRIAL: NCT07011134
Title: Effect of Early Versus Late Aminophylline Administration on Recovery Profile in Pediatric Patients Undergoing Ambulatory Surgery Under General Anesthesia; a Randomised Controlled Trial
Brief Title: Timing of Aminophylline and Recovery in Pediatric Ambulatory Surgery
Acronym: ELEAR-PAP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hany Mohammed El-Hadi Shoukat Mohammed (Other)
Responsible Party: Sponsor-Investigator, Hany Mohammed El-Hadi Shoukat Mohammed, Assistant Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MS-408-2024
Record Dates: First submitted 2025-05-12; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Recovery; Pediatric Anesthesia; Ambulatory Surgery
Keywords: pediatric; recovery of conciousness; aminophylline; sevoflurane; Ped PADSS; home readiness
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group E will receive aminophylline at an early intraoperative time immediately after fixation of E (Active Comparator): Group E (n=20): patients will receive aminophylline (5 mg/Kg) at an early intraoperative time immediately after fixation of ETT and confirmation of bilateral adequate lung ventilation (EtSevo< 1).
  Interventions: Drug: Group (E): receive aminophylline early intraoperatively,
- Group L will receive aminophylline at late intraoperative time immediately after disco (Active Comparator): Group L (n=20): patients will receive aminophylline (5 mg/Kg) at late intraoperative time immediately after discontinuation of sevoflurane (EtSevo < 1)
  Interventions: Drug: Group (L) received aminophylline late intraoperatively
- Group (C) will receive normal saline immediately after discontinuation of sevoflurane (Placebo Comparator): Group (C) (n=20): patients will receive normal saline immediately after discontinuation of sevoflurane (EtSevo < 1).
  Interventions: Drug: Group (C) will receive normal saline post-anesthetic discontinuation.

INTERVENTIONS:
Drug: Group (E): receive aminophylline early intraoperatively, — Group E (n=20): patients received aminophylline at an early intraoperative time immediately after fixation of ETT and confirmation of bilateral adequate lung ventilation (EtSevo< 1)
  Other Names: Early aminophylline group
  Arms: Group E will receive aminophylline at an early intraoperative time immediately after fixation of E
Drug: Group (L) received aminophylline late intraoperatively — Group L (n=20): patients received aminophylline at late intraoperative time immediately after discontinuation of sevoflurane (EtSevo < 1).
  Arms: Group L will receive aminophylline at late intraoperative time immediately after disco
Drug: Group (C) will receive normal saline post-anesthetic discontinuation. — Group (C) (n=20): patients received normal saline immediately after discontinuation of sevoflurane (EtSevo < 1).
  Arms: Group (C) will receive normal saline immediately after discontinuation of sevoflurane

SUMMARY:
Beyond its established use as a bronchodilator and therapy for apnea of prematurity, aminophylline has demonstrated utility in reversing the effects of anesthetics, enhancing recovery by accelerating respiratory and cognitive functions. Variations in dosage (1-6 mg/kg) have been explored, but questions persist regarding optimal timing and dosing for pediatric surgical populations to achieve maximal efficacy with minimal adverse effects.

This randomized controlled study aims to evaluate the effect of early versus late aminophylline administration on recovery profiles in pediatric patients undergoing ambulatory surgery under sevoflurane anesthesia.

Sixty children aged 4-12 years will be randomly allocated into three groups: Group (E) will receive aminophylline early intraoperatively, Group (L) will receive aminophylline late intraoperatively, and Group (C) will receive normal saline post-anesthetic discontinuation.

DETAILED DESCRIPTION:
An online randomization program (http://www. Randomizer.org) will be used to generate a random list and each patient's code will be kept in an opaque sealed envelope. Patients will be randomly allocated with 1:1:1 allocation ratio into three equal groups in a parallel manner:

* Group E (n=20): patients will receive aminophylline at an early intraoperative time immediately after fixation of ETT and confirmation of bilateral adequate lung ventilation (EtSevo< 1).
* Group L (n=20): patients will receive aminophylline at late intraoperative time immediately after discontinuation of sevoflurane (EtSevo < 1).
* Group (C) (n=20): patients will receive normal saline immediately after discontinuation of sevoflurane (EtSevo < 1). Patients and outcome assessors will be blinded to the group of the patients. An independant anesthetist who is not involved in the study will prepare the interventional medications.

Preoxygenation with 100% oxygen will be done for 3 min. An intravenous cannula will be inserted after inhalational induction of sevoflurane at 8%. Then, General anesthesia will be induced by propofol (2.0 mg/kg), fentanyl (1.0 mcg/kg) and atracurium (0.5 mg/kg) endotracheal intubation will be performed after full relaxation.

Anesthesia will be maintained with sevoflurane (2.0%-3.0%) to keep EtSevo 2.0 % in an O2/air mixture, and top up doses of atracurium every 30 min. Fresh gas flow will be set at 3 L/min all through the intraoperative period. Minute ventilation will be adjusted to maintain normocapnia (end tidal carbon dioxide; et CO2, between 32- and 34-mm Hg application of 5.0 mmHg of PEEP).

Two syringes will be prepared by an independent anesthesiologist for each patient. One syringe contains 5.0 mg/kg aminophylline while the other syringe contains a similar volume of normal saline. Then according to the allocated group, the independent anesthesiologist injected the syringe in an appropriate time and rate (over 10 min). All patients will receive Lactated Ringer's solution infused at a rate of 2.0-3.0 mL/kg/h and dexamethasone at 0.15 mg/Kg as antiemetic. Normothermia will be maintained by warming the IV fluids and using Bair Hugger warming system.

In case of tachycardia (20% increase in the heart rate from the baseline reading) or hypertension (20% increase in the mean arterial pressure from the baseline reading), the depth of anesthesia will be increased by increasing the concentration of sevoflurane and administration of IV fentanyl at 1μg/Kg. In case of hypotension (20% decrease in the mean arterial pressure from the baseline reading); if fluid boluses failed to restore blood pressure back to normal the concentration of the sevoflurane will be reduced, and ephedrine will be administered in 5.0 mg/kg increments.

In the post-anesthesia care unit (PACU), the patient will be assessed immediately after admission and every 5 min using the Pediatric Post-Anesthetic Discharge Scoring System (Ped-PADSS) until it reaches at least 9 points; then the patient will be ready to discharge home. All patients will be given 0.5 mg/Kg I.V. boluses of pethidine if pain score ( Wong-baker faces pain scale) > 4. Ramsay sedation scale will be recorded to distinguish 3 levels of sedation, where 0 means no sedation, 2-3 means conscious sedation, and 4-6 means deep sedation. Emergence delirium (ED) will be suspected if the child had a non-purposeful movement, seemed disorientated or confused, failed to interact normally with parents or caregiver or pulling IV lines, wound dressings or monitors. The Watcha scale will be used to assess postoperative emergence delirium (ED) in the recovery room. Diagnosis of ED will be considered if the child had a score of >2 on the Watcha score.

Measurement tools:

* Demographic data (age, sex, weight), ASA physical status (I or II), type and duration of surgery (from skin incision utill completion of last stitch) and duration of anaesthesia (from iv induction utill sevoflurane discontinuation).
* Heart rate (HR) and mean arterial blood pressure (MBP) will monitored continuously and recorded at the following intervals: T0= immediately before I.V. induction of GA, T1= immediately after fixation of ETT (corresponding to the start time of drug administration in group E), T3= 15 min after fixation of ETT, T4= immediately before sevoflurane discontinuation, T5= 5 min after discontinuation of sevoflurane (corresponding to the ending time of drug administration in groups L and C, T6= 5 min after extubation, T7= 10 min after transfer to PACU.
* Ramsay sedation scale will be recorded 5 min after extubation, on admission to the PACU, and when the Pediatric Post-Anesthetic Discharge Scoring System (Ped-PADSS) >9.
* Watcha scale to diagnose ED will be assessed 5min after PACU admission. ED will be considered if the child had a score of >2 after being suspected clinically and before giving the rescue analgesics.
* Pediatric Post-Anesthetic Discharge Scoring System (Ped-PADSS) will be assessed and recorded immediately after PACU admission and every 5 min until it reached at least 9 points. Recovery of consciousness (ROC) time: defined as the time interval in minutes from discontinuation of sevoflurane anesthetic to eye opening in response to verbal or tactile command (extubation criteria).
* Home readiness discharge time: which is the time in minutes taken to home discharge decision; started from admission to PACU utill Ped PADSS reached at least 9.
* Total recovery time: which is the time in minutes started from discontinuation of sevoflurane anesthesia utill Ped-PADSS reached at least 9. Outcomes

Primary outcome:

• Recovery of consciousness (ROC) time was defined as the time interval in minutes from discontinuation of anesthetics to eye opening in response to verbal command or tactile stimulation.

Secondary outcome:

* Home readiness discharge time: which is the time in minutes taken to home discharge decision; started from admission to PACU utill Ped PADSS reached at least 9.
* Total recovery time: which is the time in minutes started from discontinuation of sevoflurane anesthesia utill Ped-PADSS reached at least 9.
* Level of sedation as assessed by Ramsay sedation scale 5 min after extubation, on admission to the PACU, and when the Pediatric Post Anesthetic Discharge Scoring System (Ped-PADSS).
* Incidence of ED as assessed by Watcha scale 5 min after PACU admission. Adverse events after aminophylline administration (e.g., arrhythmia, hypotension or hypertension, tremors, seizures, vomiting, shivering, agitation, rhabdomyolysis).

Ethical consideration:

Informed consent will be obtained from all parents involved in the study. There were adequate provisions to maintain the privacy of participants and confidentiality of the data.

Sample size calculation:

The sample size calculation was performed using G.power 3.1.9.2 (Universitat Kiel, Germany). The sample size was calculated based on the following considerations: 0.05 α error and 95% power of the study to demonstrate a 10% decrease in ROC (the primary outcome) with group E than group L (mean 4.53 min and SD 3.33 min, the mean was 8.93 min and SD was 0.92 min in group C according to a previous study). Two cases were added to each group to overcome dropout. Therefore, 20 patients were allocated in each group. Statistical analysis Statistical analysis will be done by SPSS v27 (IBM©, Chicago, IL, USA). The Shapiro-Wilks test and histograms will be used to evaluate the normality of the distribution of data. Quantitative parametric data will be presented as mean and standard deviation (SD) and will be analyzed by ANOVA (F) test with post hoc test (Tukey). Quantitative non-parametric data will be presented as median and interquartile range (IQR) and will be analyzed by Kruskal-Wallis test with Mann Whitney-test to compare each group. Qualitative variables will be presented as frequency and percentage and will be analyzed utilizing the Chi-square test. A two tailed P value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age from 4 to 12 years.

  * Both sexes.
  * American society of Anesthesiologist (ASA) physical status I-II.
  * Scheduled for pediatric ambulatory elective surgical procedures lasting ≤ three hours duration.

Exclusion Criteria:

* Parents refusal to participate.

  * Conditions and diseases interfering with ambulatory day case surgery e.g., significant respiratory diseases, morbid obesity, obstructive sleep apnea, sickle cell anemia, prematurity, D.M, and family history of malignant hyperthermia.
  * Laparoscopic, endoscopic or abdominal surgeries.
  * History of cardiac arrhythmia or palpitation.
  * Patients with congenital heart, significant cardiovascular, respiratory diseases, renal impairment, hepatic dysfunction, hypo/hyperthyroidism or active peptic ulcer disease.
  * Patients with neurological, psychiatric diseases, cognitive dysfunction, epilepsy or history of convulsions.
  * Current treatment with xanthines or patient received aminophylline in the previous 24 hr. Hypersensitivity to aminophylline or other methylxanthines.
  * Patients who need alteration in the sevoflurane concentration due to either hypo/hypertension were excluded from the study and replaced.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Recovery of consciousness (ROC) time | from discontinuation of anesthetics to eye opening in response to verbal or tactile command up to 30 minutes from discontinuation of anesthetics
  Recovery of consciousness (ROC) time will be defined as the postoperative time interval in minutes from discontinuation of anesthetics to eye opening in response to verbal or tactile command up to 30 minutes from discontinuation of anesthetics.

SECONDARY OUTCOMES:
Home readiness discharge time | started from admission to PACU untill Ped PADSS reached at least 9 up to 2 hours postoperatively
  the postoperative time in minutes taken to home discharge decision; started from admission to PACU untill Ped PADSS reached at least 9 up to 2 hours postoperatively.
Total recovery time | started from discontinuation of sevoflurane anesthesia till Ped-PADSS reached at least 9 up to 2.5 hours after discontinuation of anesthetics
  the postoperative time in minutes started from discontinuation of sevoflurane anesthesia till Ped-PADSS reached at least 9 up to 2.5 hours after discontinuation of anesthetics.
Level of sedation | 5 minutes after extubation, on admission to the PACU, and when the Pediatric Post Anesthetic Discharge Scoring System (Ped-PADSS) reached 9.
  postoperatively assessed by Ramsay sedation scale at 5 minutes after extubation, on admission to the PACU, and when the Pediatric Post Anesthetic Discharge Scoring System (Ped-PADSS) reached 9. Ramsay scale distinguishes 3 levels of sedation, where 0 means no sedation, 2-3 means conscious sedation, and 4-6 means deep sedation.
Incidence of ED | 5 minutes after PACU admission.
  assessed by Watcha scale 5 minutes after PACU admission. Emergence delirium (ED) is suspected if the child has a non-purposeful movement, seemed disorientated or confused, fail to interact normally with parents or caregiver or pulling iv lines, wound dressings or monitors. The Watcha scale will be used to assess postoperative emergence delirium (ED) in the recovery room. Diagnosis of ED will be considered if the child has a score of >2 on the Watcha score.
Adverse events | postoperatively
  Postoperative adverse events after aminophylline administration (e.g., arrhythmia, hypotension or hypertension, tremors, seizures, vomiting, shivering, agitation, rhabdomyolysis) will be documented up to 2 hours postoperatively
Pediatric Post-Anesthetic Discharge Scoring System (Ped-PADSS) | immediately after PACU admission and every 5 minutes until it reached at least 9 points.
  will be assessed postoperatively and recorded immediately after PACU admission and every 5 minutes until it reached at least 9 points up to 2 hours postoperatively.

OTHER OUTCOMES:
Demographic data and clinical characteristics | preoperative assessment
  age in years
hemodynamics (1) | T0=immediately before GA induction,T1=immediately after ETT fixation,T3=15 minutes after ETT fixation,T4=immediately before sevoflurane discontinuation,T5=5 minutes after itsdiscontinuation,T6=5 minutes after extubation,T7=10 minutes after PACU transfer
  Heart rate (HR) will monitored continuously and recorded at spicified intervals
Demographic data and clinical characteristics (2) | preoperative assessment
  sex
Demographic data and clinical characteristics (3) | preoperative assessment
  weight in Kilograms
Demographic data and clinical characteristics (4) | preoperative assessment
  ASA physical status (I or II)
Demographic data and clinical characteristics (5) | preoperative assessment
  type and duration of surgery (from skin incision till completion of last stitch)
Demographic data and clinical characteristics (6) | perioperative assessment
  duration of anaesthesia (from iv induction till sevoflurane discontinuation).
hemodynamics (2) | T0=immediately before GA induction,T1=immediately after ETT fixation,T3=15 minutes after ETT fixation,T4=immediately before sevoflurane discontinuation,T5=5 minutes after itsdiscontinuation,T6=5 minutes after extubation,T7=10 minutes after PACU transfer
  mean arterial blood pressure (MBP) will monitored continuously and recorded at specified intervals

CONTACTS AND LOCATIONS:
Overall Officials: Neven AbdElmalk Gouda, MD, Study Chair — kasr Alainy Medical School/Cairo University; Menna T'Allah A.Mahmoud Gebril, MSc, Principal Investigator — kasr Alainy Medical School/Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
To help other researchers to benefit from the results

REFERENCES:
- [Background] El Tahan MR. Effects of aminophylline on cognitive recovery after sevoflurane anesthesia. J Anesth. 2011 Oct;25(5):648-56. doi: 10.1007/s00540-011-1190-8. Epub 2011 Jul 14. PMID 21755342
- [Background] Chen Yang, Tingting Wu, Linrui Tang, Xuebing Zhang. A prospective observational study comparing the pediatric post anesthesia discharge scoring system with clinical discharge criteria in pediatric day surgical patients in Western China. Research square 2012.
- [Background] Kasim SA, Bahr MH, Abdelkader M, Rashwan DAE. The effect of preoperative aminophylline on the recovery profile after major pelvic-abdominal surgeries: a randomized controlled double-blinded study. BMC Anesthesiol. 2021 Apr 19;21(1):122. doi: 10.1186/s12871-021-01340-7. PMID 33874898